CLINICAL TRIAL: NCT06279299
Title: Lateral Pelvic Lymph Node Dissection for Rectal Neuroendocrine Neoplasms Undergoing Laparoscopic Total Mesenteric Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Haitao Zhou, Clinical Professor, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLND
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Rectal Neuroendocrine Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lateral Pelvic lymph node dissection (Experimental): After performing TME surgery, further conduct lateral pelvic lymph nodes dissection.
  Interventions: Procedure: lateral pelvic lymph node dissection

INTERVENTIONS:
Procedure: lateral pelvic lymph node dissection — Following the total mesorectal excision principle, the rectum and mesentery are removed, with careful protection of the pelvic autonomic nerves. After completing laparoscopic rectal resection, lateral lymph node dissection is performed. The lateral dissection follows these steps: ① Open the peritoneum at the bifurcation of the iliac vessels, dissect along the retroperitoneum adjacent to the ureter-bladder fascia, expose the lateral pelvic area, and carefully protect the ureter and hypogastric nerves. Open the peritoneum along the edge of the external iliac vessels close to the inguinal ligament, clear the lymphatic fatty tissue alongside the external iliac vessels along the edge of the iliopsoas and internal oblique muscles; ② After identifying the hypogastric nerve, dissect along the bladder-bladder fascia, separate the bladder and the fat tissue around the lateral pelvic space, completely remove the lymphatic tissue around the internal iliac vessels and hypogastric nerves.

SUMMARY:
The purpose of this study is to investigate the metastatic status of lateral pelvic lymph nodes in rectal neuroendocrine neoplasms (rNENs) undergoing laparoscopic total mesenteric excision (TME). The hypothesis is that the rate of lateral lymph node metastasis is underestimated in rNENs undergoing TME, necessitating concurrent lateral Pelvic lymph node dissection.

DETAILED DESCRIPTION:
This study is a prospective single-arm clinical study. 30 patients with rNENs undergoing TME are planned to be included in the study. The purpose of this study is to investigate the metastatic status of lateral pelvic lymph nodes in (rNENs) undergoing laparoscopic TME. The primary endpoint is the rate of lateral pelvic lymph nodes metastasis. The primary hypothesis was the rate of lateral lymph node metastasis is underestimated in rNENs undergoing TME, necessitating concurrent lateral Pelvic lymph node dissection.

This study seeks to report for the first time the true status of lateral pelvic lymph node metastasis in these patients. In addition, the proportion of patients with radical resection (R0), surgical complication profile, and quality of life (QoL) are also secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven rectal neuroendocrine neoplasm (neuroendocrine tumor and carcinoma);
2. Meets any one of the following conditions:

   * Preoperative imaging examinations reveal that the maximum diameter of the tumor is greater than 2cm.
   * Preoperative imaging examinations reveal that the maximum diameter of the tumor is between 1-2cm and the clinical staging is T2 or higher.
   * Preoperative imaging examinations reveal that the maximum diameter of the tumor is between 1-2cm and is categorized as Grade 3 differentiation.
   * Recurrence after local excision under endoscopy.
3. Eastern Cooperative Oncology Group(ECOG) performance score ≤ 1;
4. Written informed consent;

Exclusion Criteria:

1. Complete intestinal obstruction;
2. Hepatitis activity and peripheral neuropathy (such as peripheral neuritis, pseudo meningitis, motor neuritis, and sensory impairment);
3. Significant organ dysfunction or other significant diseases, including clinically relevant coronary artery disease, cardiovascular disease, or myocardial infarction within the 12 months before enrollment; severe neurological or psychiatric history; severe infection; active disseminated intravascular coagulation；
4. Pregnancy or breastfeeding;
5. Alcohol abuse or drug addiction;
6. Concurrent uncontrolled medical condition;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of lateral pelvic lymph node metastasis | up to 14 days
  The rate of lateral pelvic lymph node metastasis = lateral pelvic lymph node metastasis cases/all cases.

SECONDARY OUTCOMES:
The rate of lymph node metastasis | up to 14 days
  The rate of lymph node metastasis = lymph node metastasis cases/all cases.
Disease-free survival rate | three years
  Disease-free survival (DFS) is a number that tells the chances of staying free of a disease or cancer after a particular treatment. It is the percentage of individuals in the treatment group who are likely to be free of the signs and symptoms of a disease after a specified duration of time.
Overall survival rate | three years
  The time from diagnosis to (for any reason) death.
Locoregional recurrence free survival rate | three year
  Locoregional Recurrence Free Survival is defined as the time interval between the day of diagnosis in the study and the date of local relapse/recurrence or regional relapse/recurrence whichever occurs first.
Radical resection (R0) | up to 14 years
  R0 resection rate is R0 resection probability of radical surgery in patients with locally advanced rectal cancer after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhou, Study Chair — National Cancer Center, China
Locations (1):
- National Cancer Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Participants' data are only allowed to be used for the analysis of this study and are not authorized to be shared with other researchers.